CLINICAL TRIAL: NCT00709332
Title: An Open-label Pharmacokinetic Drug Interaction Study of Folic Acid and 250 Mcg NGM/35 Mcg E E (ORTHO-CYCLEN) in Healthy Women.
Brief Title: A Drug Interaction Study of Folic Acid and Oral Contraceptive Tablets Containing Norgestimate (NGM)/Ethinyl Estradiol (EE) in Healthy Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR002206
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Drug Interactions; Contraception; Pharmacokinetics
Keywords: Norgestimate; Folic Acid; Ortho-Cyclen; Female contraception; Ethinyl Estradiol; Drug Interactions; Pharmacokinetics; Contraceptives, Oral
MeSH Terms: interventions — norgestimate; Ethinyl Estradiol; Folic Acid

INTERVENTIONS:
Drug: Norgestimate; Ethinyl Estradiol; Folic acid

SUMMARY:
The purpose of the study is to assess the effect of folic acid administration on the blood level and the breakdown products of oral contraceptive (OC) [250 mcg NGM/35 mcg EE] tablets.

DETAILED DESCRIPTION:
This is an open-label, randomized (study drug assigned by chance), single-center, pharmacokinetic interaction study. Healthy adult women who met the prestudy eligibility criteria were randomized to 1 of 2 treatment groups. The randomization was balanced using permuted blocks. Healthy volunteers in Group 1 were to receive a single oral dose of 250 µg NGM/35 mcg EE (1 tablet) on Days 1 and 17, and 1 mg of folic acid on Days 4 through 18. Healthy volunteers in Group 2 were to receive a single, oral 1 mg dose of folic acid on Days 1 and 17, and 1 tablet on Days 2 through 17. Serial blood samples were to be collected from each healthy volunteer on Days 1 and 17 before dosing and at specified times for up to 72 hours after dosing for pharmacokinetic evaluation. Healthy volunteers were to be confined overnight at the study unit on Days -1 and 16 for an overnight fast of at least 8 hours before dosing on Days 1 and 17. Healthy volunteers were to remain confined at the study unit until the 24-hour blood samples were collected on Days 2 and 18. Safety was based on the incidence of adverse events, and on changes in clinical laboratory values, vital signs, electrocardiograms, and physical and gynecological examination findings. The Sponsor prematurely terminated this study on 14 February 2005 because of errors made at the study site in healthy volunteer randomization, the timing of blood draws, and handling of laboratory samples. As a result of these errors, the pharmacokinetic samples collected were not analyzed, and a new study was initiated (NRGMON-CON-1006). Due to the premature termination of the study, no healthy volunteer received more than 9 days of therapy. Most healthy volunteers completed the screening and premature termination procedures.

Oral contraceptives tablet (250 mcg NGM/35 mcg EE); Folic acid tablet (1 mg). Group 1: Single OC tablet on Days 1 and 17, 1 folic acid tablet on Days 4 to 18. Group 2: Single folic acid tablet on Days 1 and 17, 1 OC tablet on Days 2 to 17. The study drugs were to be taken with 240 mL (8 oz) of water at approximately 8:00 a.m. Healthy volunteers were required to fast for a minimum of 8 hours before dosing on Days 1 and 17.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Nonpregnant
* Nonlactating
* Nonsmoking women
* Weighing at least 110 pounds
* With regular menstrual cycles
* A body mass index between 16 and 29.9 kg/m2
* And a hematocrit of at least 36%

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to sex hormonal therapy including: thromboembolic disorders cerebral vascular or coronary artery disease, chronic untreated hypertension, or migraines, benign or malignant liver tumor that developed during the use of OC
* Known or suspected estrogen-dependent neoplasia
* Presence of disorders commonly accepted as contraindications to combined OC including: undiagnosed abnormal vaginal bleeding, any neurovascular lesion of the eye or serious visual disturbance, or liver disease
* Intake any multivitamin or folic acid-containing supplements within 30 days before study admission
* Used a steroid hormone-containing intrauterine device within 3 months prior to study admission
* Used any medications that were known cytochrome P-450 enzyme inducers or inhibitors (e.g., St. John's Wort, cimetidine or rifampin), within 60 days before dosing.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2005-01; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetic drug interaction between folic acid and OC (250 mcg NGM and 35 mcg EE) as measured by the pharmacokinetics of the active breakdown products of NGM, (norelgestromin [NGMN], and norgestrel [NG]) and EE.

SECONDARY OUTCOMES:
Safety is also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L.C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A drug interaction study of folic acid and oral contraceptive tablets containing norgestimate (250 mcg)/ethinyl estradiol (35 mcg) in healthy women — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=456&filename=CR002206_CSR.pdf